CLINICAL TRIAL: NCT06596408
Title: Evaluation of Retinal Vascular Density in High Myopia Without Pathological Myopic Maculopathy Using OCTA .
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Sara Magdy Mohamed, Principal Investigator, Sohag University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: Vascular Density in high Myope
Record Dates: First submitted 2024-08-30; First posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: High Myopia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- High Myopes of spherical error -6 and more . (Experimental): About 50 participants with high myopia will undergo evaluation of their macular vascular density using OCTA and also central macular thickness using OCT.
  Interventions: Other: optical coherence tomography angiography

INTERVENTIONS:
Other: optical coherence tomography angiography — OCTA will be used to evaluate the macular vascular density and to exclude patients with pathological myopic maculopathy

SUMMARY:
Study aiming to evaluate Macular Vascular Density in High Myopes without pathological myopic maculopathy in outpatient clinic in Sohag teaching hospital using OCTA .

DETAILED DESCRIPTION:
Study Design : This is a cross sectional observational study , of about 50 patients attending ophthalmology outpatient clinic at Sohag Teaching Hospital .

Inclusion criteria :

All myopic patients with axial high myopia (-6 spherical refractive error or more) attending the ophthalmology outpatient clinic .

Exclusion criteria :

The exclusion criteria will include :

* History of other any ocular diseases , systemic diseases that may affect the ocular circulation .
* Previous intraocular surgery or ocular injury .
* Any patient with pathological myopic maculopathy (epiretinal membrane, foveoschisis, macular holes, lamellar holes, Lacquers cracks, choroidal neovascularization and retinal atrophy ) .

ELIGIBILITY:
Inclusion Criteria wil include :

* All myopic patients with axial high myopia (-6 spherical refractive error or more) of different age groups .

Exclusion Criteria will include :

* -History of other any ocular diseases , systemic diseases that may affect the ocular circulation .
* Previous intraocular surgery or ocular injury .
* Any patient with pathological myopic maculopathy as epiretinal membrane, foveoschisis, macular holes, lamellar holes, Lacquers cracks, choroidal neovascularization and retinal atrophy .

Min Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2024-09-11 (Estimated); Primary Completion 2025-09 (Estimated); Study Completion 2025-10 (Estimated)

PRIMARY OUTCOMES:
Outcome of evaluation of vascular density in high myopes | 6 month
  Correlation between macular vascular density in high myopes and their :
  Uncorrected visual acuity in diopters . Best corrected visual acuity in diopters . Spherical equivalent refraction that measured through this equivalent (spherical error + 1/2 cylindrical error ) .
  Central macular thickness in micrometers .
  To see how does ischemia affects vision in high myopes .

CONTACTS AND LOCATIONS:
Overall Officials: Adham Salah Mohammed, lecturer, Study Chair — Sohag University
Locations (1):
- Sohag University, Sohag, Sohag Governorate, Egypt

IPD SHARING:
Plan to Share IPD: Undecided